CLINICAL TRIAL: NCT03002259
Title: Evaluation of Dexamethasone in Cardiac Surgery Using a Novel Trial Design
Brief Title: Dexamethasone for Cardiac Surgery-II Trial
Acronym: DECS-II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Response
Keywords: cardiac surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No placebo required
- Dexamethasone (Active Comparator): Dexamethasone, 1 mg/kg (maximal dose 100 mg), single dose administration before cardiopulmonary bypass
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone administered as a single IV injection after induction of anaesthesia, but before initiation of CPB. Prepare as a 20 mg/mL dexamethasone solution, made up with 0.9% saline to 10 ml.
  Arms: Dexamethasone

SUMMARY:
Background. Numerous studies have investigated high-dose corticosteroids in cardiac surgery, but with mixed results leading to ongoing variations in practice around the world. The Dexamethasone for Cardiac Surgery-II Trial (DECS-II) is a study comparing high-dose dexamethasone with placebo in patients undergoing cardiac surgery.

Methods. We discuss the rationale for conducting DECS-II, a 2800-patient, pragmatic, multicenter, assessor-blinded, randomized trial in cardiac surgery, and the features of the DECS-II study design (objectives, end points, target population, balanced clusters based on practice preference with post-randomization consent, treatments, patient follow-up and analysis).

Conclusions. The DECS-II Trial will use a novel, efficient trial design to evaluate whether high-dose dexamethasone has a patient-centered benefit of enhancing recovery and increasing the number of days at home after cardiac surgery.

DETAILED DESCRIPTION:
High-dose corticosteroids attenuate the inflammatory response to surgery with CPB and are commonly used in some countries,but uncommonly in the US, Canada and Australia. Steroids can reliably attenuate activation of the complement pathways associated with cardiac surgery, but clinical trials have had mixed results. The current evidence is dominated by the results of two recent large randomized trials: DECS (n=4,494)6 and SIRS (n=7,507).

Both DECS and SIRS assigned patients undergoing cardiac surgery with CPB to receive either a high intraoperative dose of steroids (dexamethasone 1 mg/kg, or methylprednisolone 500 mg, respectively) or placebo. The point estimates of both trials suggested a possible reduction in serious complications and mortality. Planned subgroup analyses in the DECS trial steroids reduced the incidence of respiratory failure (3.0 % vs. 4.3%, P=0.02), infection (9.5% vs. 14.8%, P=0.009), and shortened hospital stay (median 8 [7-13] vs. 9 [7-13] days, P=0.009).6 Severe renal failure (need for RRT) was reduced, 0.4% vs. 1.0%, P=0.04.8 But SIRS found methylprednisolone was associated with a higher incidence of myocardial injury (as measured by elevation of CK-MB enzyme). Nether trial identified a higher risk of myocardial infarction (MI). The methylprednisolone-induced elevation of CK-MB may therefore be a class effect.

Another compelling finding in pre-planned subgroup analysis of patient age groups is that when limiting analysis to those aged less than 75 years in the DECS trial, dexamethasone reduced the risk of the primary composite endpoint, RR 0.74 (95% CI: 0.58-0.95), P=0.017; as well as respiratory failure RR 0.62 (95% CI: 0.42-0.91), P=0.014; and possibly mortality RR 0.53 (95% CI: 0.26-1.10), P=0.08.6 This age-interaction effect is supported by the demonstration of increased C-reactive protein concentrations in younger patients enrolled in the DECS trial.

Therefore, it is highly plausible that prophylactic steroids can suppress deregulated inflammation and thus improve outcomes in cardiac surgery, but only when used in a less elderly (i.e. <75 years) patient population.

In retrospect, the primary endpoints of both DECS and SIRS trials can be challenged, in that they used composites heavily weighted by thrombotic events (MI, stroke) and not specific to inflammation (respiratory failure, kidney injury, sepsis, prolonged ICU and hospital stay, mortality). We thus plan to re-evaluate dexamethasone in cardiac surgery, using a patient-centred, clinically important endpoint focused on enhanced recovery and earlier hospital discharge: "days alive and at home up to 30 days after surgery".

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 18 to 75 years undergoing elective cardiac surgery with cardiopulmonary bypass
2. EuroScore-II estimated risk of 1.5% or higher

Exclusion Criteria:

1. Poor language (English or Dutch) comprehension
2. Type I diabetes
3. Endocarditis or other evidence of sepsis
4. Preoperative steroid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1956 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
days at home up to 30 days after surgery | 30 days from Start of Surgery
  Home is defined as a person's usual abode or that of a close relative, excluding any nursing facility (rehabilitation center or nursing home).

SECONDARY OUTCOMES:
respiratory failure | 30 days from Start of Surgery
  Uninterrupted postoperative mechanical ventilation for more than 48 hours from admission to ICU
Infection | 30 days from Start of Surgery
  Surgical site infection, pneumonia, or documented positive microbial culture from any site (including blood).
Myocardial Infarction | 30 days from Start of Surgery
  Postoperative myocardial infarction will be defined according to the third universal definition
Stroke | 30 days from Start of Surgery
  A new neurological deficit lasting more than 24 hours or leading to earlier death, and confirmed by medical imaging.
Peak blood glucose | 30 days from Start of Surgery
  The highest blood glucose measured in this same period
Length of stay | 30 days from Start of Surgery
  Time from postoperative ICU admission to ICU discharge (hours) and hospital discharge (days).
Quick SOFA score | Each evening on days 1-3 after surgery
  Tachypnoea, altered mentation and/or hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, MBBS, MD, Principal Investigator — Alfred Hospital, Monash University
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbasciano RG, Olivieri GM, Chubsey R, Gatta F, Tyson N, Easwarakumar K, Fudulu DP, Marsico R, Kofler M, Elshafie G, Lai F, Loubani M, Kendall S, Zakkar M, Murphy GJ. Prophylactic corticosteroids for cardiopulmonary bypass in adult cardiac surgery. Cochrane Database Syst Rev. 2024 Mar 20;3(3):CD005566. doi: 10.1002/14651858.CD005566.pub4. PMID 38506343
- [Derived] Myles PS, Dieleman JM, Forbes A, Heritier S, Smith JA. Dexamethasone for Cardiac Surgery trial (DECS-II): Rationale and a novel, practice preference-randomized consent design. Am Heart J. 2018 Oct;204:52-57. doi: 10.1016/j.ahj.2018.06.008. Epub 2018 Jun 21. PMID 30081275